CLINICAL TRIAL: NCT04077736
Title: A Pilot Study of Low Dose IL-2 in the Treatment of Relapsing Polychondritis
Brief Title: Low-dose Recombinant Human IL-2 for the Treatment of Relapsing Polychondritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, HeJing, Proffesor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019PHB089-02
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Relapsing Polychondritis
Keywords: Relapsing polychondritis，IL-2
MeSH Terms: conditions — Polychondritis, Relapsing | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interleukin-2 (Experimental): low dose interleukin-2 injected subcutaneously, at a dose of 1 million IU five days per week for 4 weeks (day1-5, 8-12, 15-19, 22-26) and then once a week for 8 weeks (day33, 40, 47, 54, 61, 68, 75, 82).
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — low dose interleukin-2 injected subcutaneously, at a dose of 1 million IU five days per week for 4 weeks (day1-5, 8-12, 15-19, 22-26) and then once a week for 8 weeks (day33, 40, 47, 54, 61, 68, 75, 82).
  Other Names: Recombinant Human Interleukin-2

SUMMARY:
Relapsing polychondritis (RP) is a rare, systemic autoimmune disorder characterized by episodic inflammation of cartilaginous structures. Pro-inflammatory chemokines involved in the recruitment of monocytes and modulation of macrophage function, such as monocyte chemoattractant protein-1, macrophage inflammatory protein 1β, and interleukin (IL)-8, are significantly elevated in active RP compared with controls.The activation of monocytes and macrophages may play an important role in the pathophysiology of RP. The levels of serum Th1 cytokines (interferon, IL-2 (IL-2) and IL-12 (IL-12) were significantly correlated with disease status，which suggested that RP may be a Th1-mediated disease process. IL-2 is a kind of lymphocyte growth factor. At lower doses, regulatory T cells exhibit dominant amplification because of their more sensitivity to IL-2. Regulatory T cells can inhibit the growth of effector T cells and then play an immunosuppressive role. The investigators hypothesized that low-dose IL-2 could be a novel therapy in active RP patients. This clinical study will explore the efficacy and immunological evaluation of low dose IL-2 in the treatment of RP.

DETAILED DESCRIPTION:
Ten patients with active RP at 18 to 70 years of age were enrolled. Without changing the original treatment plan, IL-2 1 million units was administered subcutaneously five days every week for 4 weeks and then once a week for 8 weeks. The clinical symptoms, disease score scale, laboratory parameters, immune cell subsets and cytokines should be monitored during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 and ≤70 years
2. Meet the revised Michet criteria
3. Patients had an inadequate response to standard treatment for ≥ 4 weeks. The background treatment included corticosteroids (≤0.5 mg/ kg), immunosuppressants ( methotrexate, hydroxychloroquine, azathioprine, mycophenolate mofetil leflunomide, or cyclophosphamide)
4. Negative urine pregnancy test
5. Written informed consent form

Exclusion Criteria:

* Any subject who meets any of the following criteria shall be excluded:

  1. Use rituximab or other monoclonal antibodies within 1.6 months.
  2. 1 months after treatment with high dose glucocorticoid (> 1 mg/kg/d).
  3. Serious complications: heart failure (≥ New York Heart Association（NYHA） III grade), renal insufficiency (creatinine clearance rate ≤ 30 ml/min), liver function insufficiency (serum alanine transaminase or glutamic-pyruvic transaminaseT > 3 times normal upper limit, or total bilirubin > normal upper limit)
  4. Other serious, progressive or uncontrollable hematological, gastrointestinal, endocrine, lung, heart, nerve, or brain diseases (including demyelination diseases, such as multiple sclerosis).
  5. Known allergies, hyperresponsiveness or IL-2 or its excipients are intolerant.
  6. Severe infections (including, but not limited to, hepatitis, pneumonia, bacteremia, pyelonephritis, Epstein-Barr virus, tuberculosis infection), hospitalization for infection, or intravenous antibiotics 2 months before the first dose of treatment.
  7. Chest imaging showed abnormalities in malignant tumors or current active infections (including tuberculosis) within 3 months before the first use of the study.
  8. Infected with HIV (HIV antibody positive serology) or hepatitis C (Hep C antibody positive serology). If seropositive, consult a doctor with expertise in the treatment of HIV or hepatitis C virus infection.
  9. There has been any known malignant tumor or history of malignant tumor in the past 5 years (with the exception of non-melanoma skin cancer, non-melanoma skin cancer with no sign of recurrence or surgically cured cervical tumor within 3 months of use of the first study preparation).
  10. There are uncontrolled mental or emotional disorders, including a history of drug and alcohol abuse over the past three years, which may hinder the successful completion of the study.
  11. Within 3 months before the first injection of the research agent, during the study period or within 4 months after the last injection of the research agent, any live virus or bacterial vaccine is received or expected to be received. Bacillus Calmette-Guerin was vaccinated within 12 months after screening.
  12. Pregnant and lactating women (WCBP) are reluctant to use medically approved contraceptives during and 12 months after treatment.
  13. Men whose partners have fertility potential but do not want to use appropriate medically approved contraceptives during and within 12 months of treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Foxp3+Treg cells: change in percentage of total lymphocytes | week 12
  Treg refers to regulatory T cells

SECONDARY OUTCOMES:
Relapsing Polychondritis Disease Activity Index | week 12
  Relapsing Polychondritis Disease Activity Index
safety assessment | week 12
  Adverse events includes injection site reactions, influenza-like symptoms, infection, fever, tumor,drug-induced liver and kidney damage.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhanguo, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No